CLINICAL TRIAL: NCT01956630
Title: Clinical Study of Genetically Modified Dendritic Cells Combining to Cytokine-Induced Killer Cells for Patients With Relapse Acute Leukemia After Allo-HSCT
Brief Title: Clinical Study of DC Plus CIK for Patients With Relapse Acute Leukemia After Allo-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-DC/CIK-Leukemia
Record Dates: First submitted 2013-09-23; First posted 2013-10-08 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genetically modified DCs plus CIK cells (Experimental): Patients received four subcutaneous injections of 2-5×10e7 cells of DCs at the groin, axilla, and neck respectively on days 7, 9, 11, and 13 and i.v. infusions of 2-15×10e9 CIK on days 11 and 13 per cycle. The cycle was repeated until Wilms' tumor 1(WT1) turned negative by polymerase chain reaction(PCR) or graft-versus-host disease(GVHD) appeared.
  Interventions: Biological: Genetically modified DCs plus CIK cells
- Donor leukocyte infusions (DLI) (Active Comparator): Patients received DLI at a dose of 2×10e7/kg, 5×10e7/kg and 1×10e8/kg cluster of differentiation 3(CD3)+ cells at months 1, 2 and 3 respectively unless GVHD appeared.
  Interventions: Biological: Donor leukocyte infusions (DLI)

INTERVENTIONS:
Biological: Genetically modified DCs plus CIK cells
  Arms: Genetically modified DCs plus CIK cells
Biological: Donor leukocyte infusions (DLI)
  Arms: Donor leukocyte infusions (DLI)

SUMMARY:
Allogeneic hematopoietic cell transplantation(Allo-HSCT) is currently an effective treatment for Acute leukemia (AL). Relapse after transplantation, being a main obstacle for patient survival, is so far treated by second transplantation and donor leukocyte infusion (DLI), which seems to have high risk and low survival. Need for a new medication on relapse is urgent. The immunotherapy using Dendritic cells (DCs) combined with cytokine induced killer (CIK) cells holds promise for the adjuvant treatment of AL to eradicate or control residual disease. This randomized study was conducted to evaluate the feasibility and effective of genetically modified DCs combining to CIK immunotherapy in relapse AL after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* AL patients according to the WHO criteria
* expected survival duration of more than 3 months
* age between 8 and 61years

Exclusion Criteria:

* underlying autoimmune disease
* positive serology for HIV infection
* chronic active hepatitis

Ages: 8 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 3 years

SECONDARY OUTCOMES:
Gvhd incidence | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, Doctor, Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, China

REFERENCES:
- [Derived] Wang D, Huang XF, Hong B, Song XT, Hu L, Jiang M, Zhang B, Ning H, Li Y, Xu C, Lou X, Li B, Yu Z, Hu J, Chen J, Yang F, Gao H, Ding G, Liao L, Rollins L, Jones L, Chen SY, Chen H. Efficacy of intracellular immune checkpoint-silenced DC vaccine. JCI Insight. 2018 Feb 8;3(3):e98368. doi: 10.1172/jci.insight.98368. eCollection 2018 Feb 8. PMID 29415891